CLINICAL TRIAL: NCT00514839
Title: Brief Intervention for Regular Prescription Drug Use and Prescription Drug Use Disorders in General Hospital
Brief Title: Brief Intervention for Prescription Drug Misuse in General Hospital
Acronym: MIMIK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Luebeck (Other)
Collaborators: Federal Ministry of Health, Germany (Other Government)
Responsible Party: Principal Investigator, Hans-Jürgen Rumpf, PD Dr. Hans-Jürgen Rumpf, University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 150268661
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Substance-related Disorders
Keywords: Prescription drug use disorder; Brief intervention; General hospital; Motivational Interviewing
MeSH Terms: conditions — Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C (No Intervention): Control group receiving a booklet on health behavior
- MI (Experimental): Counselling based on Motivational Interviewing plus individualized feedback
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Motivational Interviewing — Two sessions of Motivational Interviewing (after baseline assessment and 4 weeks later) plus one individualized feedback based on the Transtheoretical Model of Behavior Change (8 weeks after baseline assessment)
  Arms: MI

SUMMARY:
In a randomized controlled trial, patients recruited in a general hospital and fulfilling criteria for regular consumption (more than 60 days within the last three months), dependence or abuse of prescription drugs will be randomly allocated to two conditions:(1) Intervention group consisting of two counselling sessions based on Motivational Interviewing plus a personalized feedback, (2) Control group receiving a booklet on health behavior.

Outcome assessment will be conducted after 12 months. The hypothesis is that counseling leads to greater reduction in consumption of prescription drugs (including discontinuation) and elevated readiness to change at follow-up.

DETAILED DESCRIPTION:
Background: Dependence on prescription drugs (DPD) is highly prevalent, whereby rate of substance specific treatment is low. A pilot study revealed elevated prevalence rates in general hospital patients compared to the general population and a positive attitude of patients suffering from DPD towards counseling. Brief intervention delivered in general hospital might be useful to promote discontinuation of prescription drug use and utilization of formal help.

Objectives: To test the efficacy of a brief intervention based on Motivational Interviewing in proactively recruited general hospital patients randomly allocated to an intervention or a control group. Methods: Patients aged 18 to 69 years are proactively recruited in surgical and internal wards of two general hospitals in the northern German city of Lübeck. Patients with regular use of prescription drugs in the last three months and/or prescription drug dependence or -abuse are randomly assigned to two conditions: (1) an intervention group with two counseling sessions based on Motivational Interviewing plus one individualized feedback based on the Transtheoretical Model of behavior change (TTM) or (2) as usual care. Outcome measures are reduction or discontinuation of prescription drug use and utilization of formal help. The efficacy of the intervention will be examined within a 3 and a 12 month follow up.

Expected impact: Findings are expected to provide evidence for brief interventions for prescription drug misuse to be used in primary care. This would be the first international results confirming such an approach in the field of prescription drug misuse. If a brief interventions would be effective, this could enhance secondary prevention for this under served population. Therefore, data are of great public health interest.

ELIGIBILITY:
Inclusion Criteria:

* Prescription drug abuse
* Prescription drug dependence
* Regular prescription drug consumption (>60 times/last three months)

Exclusion Criteria:

* Current treatment for substance abuse problems
* Terminal illness

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2005-11; Primary Completion 2008-08 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Discontinuation of consumption of prescription drugs | one year
Reduction of consumption of prescription drugs | one year
Utilization of formal help | one year

SECONDARY OUTCOMES:
Readiness to change consumption of prescription drugs | one year

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Juergen Rumpf, Ph.D., Principal Investigator — University of Luebeck

REFERENCES:
- [Derived] Zahradnik A, Otto C, Crackau B, Lohrmann I, Bischof G, John U, Rumpf HJ. Randomized controlled trial of a brief intervention for problematic prescription drug use in non-treatment-seeking patients. Addiction. 2009 Jan;104(1):109-17. doi: 10.1111/j.1360-0443.2008.02421.x. PMID 19133895